CLINICAL TRIAL: NCT04496661
Title: Searching for the Optimal tDCS Target Combined With Peripheral Electrical Stimulation in Chronic Low Back Pain: a Protocol for a Pilot Randomized Controlled Trial
Brief Title: Searching for the Optimal tDCS Target Combined With Peripheral Electrical Stimulation in Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator and Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Painmodulation
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: PES; tDCS
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated via an online generator (www.random.org) in one of three groups (1:1:1): anodal tDCS of M1 + PES; anodal tDCS of DLPFC + PES; Sham of M1 + PES.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly allocated via an online generator (www.random.org) in one of three groups (1:1:1): anodal tDCS of M1 + PES; anodal tDCS of DLPFC + PES; Sham of M1 + PES. This sequence will be performed blindly, independently, and remotely by a blind investigator who will have no contact with other research procedures, and randomization will be hidden until the group is allocated.
  The hidden allocation process will be performed using sequential, numbered, opaque and sealed envelopes. The outcome assessors, trialists (care provider and investigator) and participants will be blinded to the performed procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS over M1 and PES (Experimental): Anodic transcranial direct current stimulation (tDCS) over right primary motor cortex (M1) and PES (20Hz and 330ms) placed at the height between the T12 and S1 vertebrae in order to cover the entire lumbar area . Duration: 30 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation on M1 and Peripheral Electrical Stimulation
- tDCS over DLPFC and PES (Experimental): Anodic transcranial direct current stimulation (tDCS) over left dorsolateral prefrontal cortex (DLPFC) and PES (20Hz and 330ms) placed at the height between the T12 and S1 vertebrae in order to cover the entire lumbar area . Duration: 30 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation on DLPFC and Peripheral Electrical Stimulation
- Sham tDCS and PES (Sham Comparator): Sham tDCS and PES stimulation. Anodic transcranial direct current stimulation (tDCS) over right primary motor cortex (M1) and PES (20Hz and 330ms) placed at the height between the T12 and S1 vertebrae in order to cover the entire lumbar area. The currents will be turned off automatically after 30 seconds. Duration: 30 minutes.
  Interventions: Device: Sham tDCS and PES

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation on M1 and Peripheral Electrical Stimulation — Patients will be submitted to 10 treatment sessions, five days a week, for 30 minutes, paired to the same PES protocol. The participants will be positioned in ventral decubitus position. The direct current (2 mA) will be transferred through a neuro-stimulator (TransCranial Technologies, Hong Kong, China), with the use of electrodes and 4x4 cm sponges moistened with 0.9% saline solution. The anodic electrode will be placed on C3 to stimulate the left primary motor cortex according to the international 10-20 EEG system. The reference electrode will be positioned in the supra orbital contralateral region. For the PES, four self-adhesive electrodes with dimensions of 5 x 5 cm will be placed at the height between the T12 and S1 vertebrae in order to cover the entire lumbar area. A 20Hz frequency and pulse duration of 330ms will be provided by means of two channels from an electro-stimulator (Neurodyn, Ibramed).
  Arms: tDCS over M1 and PES
Device: Transcranial Direct Current Stimulation on DLPFC and Peripheral Electrical Stimulation — Patients will be submitted to 10 treatment sessions, five days a week, for 30 minutes, paired to the same PES protocol. The direct current (2 mA) will be transferred through a neuro-stimulator (TransCranial Technologies, Hong Kong, China), with the use of electrodes and 4x4 cm sponges moistened with 0.9% saline solution. The anodic electrode will be placed on F3 to stimulate the left dorsolateral cortex according to the international 10-20 EEG system. The reference electrode will be positioned in the supra orbital contralateral region. For the PES, four self-adhesive electrodes with dimensions of 5 x 5 cm will be placed at the height between the T12 and S1 vertebrae in order to cover the entire lumbar area. A 20Hz frequency and pulse duration of 330ms will be provided by means of two channels from an electro-stimulator (Neurodyn, Ibramed).
  Arms: tDCS over DLPFC and PES
Device: Sham tDCS and PES — For sham tDCS and PES stimulation, patients will be submitted to 10 treatment sessions, five days a week, for 30 minutes. The anodic electrode will be positioned on the left primary motor cortex, but the current will be turned off automatically after 30 seconds. The reference electrode will be positioned in the supra orbital contralateral region. For sham PES stimulations, four self-adhesive electrodes with dimensions of 5 x 5 cm will be placed at the height between the T12 and S1 vertebrae in order to cover the entire lumbar area. A 20Hz frequency and pulse duration of 330ms will be provided by means of two channels from an electro-stimulator (Neurodyn, Ibramed), but the current will be turned off automatically after 30 seconds.
  Arms: Sham tDCS and PES

SUMMARY:
Low back pain (LBP) has been associated with severe impairments, primarily related to activities of daily living, functional ability and quality of life. A multimodal approach to pain management, such as transcranial direct current stimulation (tDCS) and peripheral electrical stimulation (PES), may improve outcomes in chronic LBP. However, the optimal cerebral target for stimulation still remains controversial. This pilot trial aims to investigate whether active stimulation could promote additional gains to the PES results in LBP participants. The secondary objective is to investigate whether the stimulation of primary motor cortex and dorsolateral prefrontal cortex results in distinct clinical effects for the participants involved.

DETAILED DESCRIPTION:
For this, a pilot, sham-controlled, double-blind, randomized clinical trial in accordance with the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines. Sixty participants with chronic low back pain will be randomized into one of three tDCS groups associated with PES: motor primary cortex, dorsolateral prefrontal cortex and sham stimulation. Each group will receive transcranial direct current stimulation at an intensity of 2 mA for 30 minutes daily for 10 consecutive days. Participants will be assessed with a Brief Pain Inventory (BPI), Roland Morris Disability Questionnaire (RMDQ), Medical Outcomes Study 36-item Short - Form Health Survey (SF-36) and electromyography at baseline, endpoint (after 10 sessions) and 1-month follow up. This study will help to clarify the additive effects of tDCS combined with peripheral electrical stimulation on pain relief, muscle function and improvement in quality of life. Additionally, the investigators will provide data to identify optimal targets for management of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Diagnosis of chronic low back pain, lasting more than 6 months (The diagnosis of chronic lumbar pain will be based on clinical and neurophysiological criteria, according to the European Guidelines on Low Back Pain);
* Pain intensity of at least 4 in 10 in Visual Analogue Scale (VAS);
* Stable pharmacological treatment for at least one month before the study and throughout the study;

Exclusion Criteria:

* Intense pain from another origin, such as neuropathic pain;
* Alcohol or substance abuse;
* Associated diseases of the peripheral or central nervous system;
* Contraindications for non-invasive brain stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity | Baseline, endpoint (after 2 weeks) and the follow-up (after 1 month)
  Pain severity will be assessed with Numerical Rating Scales (NRS), which refers to a subjective measure in which individuals classify their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain) to 10 (worst pain imaginable).
Changes in pain interference in activities of daily living | Baseline, endpoint (after 2 weeks) and the follow-up (after 1 month)
  The Brief Pain Inventory (BPI) assesses multidimensional aspects of pain. It includes 15 items that evaluate the existence, severity, location, functional interference, applied therapeutic strategies and effectiveness of pain treatment. It is an instrument with adequate validity and reproducibility, commonly used in the evaluation of patients with chronic pain.

SECONDARY OUTCOMES:
Functional disability associated with chronic low back pain measured by Roland Morris Disability Questionnaire (RMDQ) | Baseline, endpoint (after 2 weeks) and the follow-up (after 1 month)
  The Roland Morris Disability Questionnaire (RMDQ) functional disability associated with chronic low back pain. Composed of 24 questions, with a variation of scores between 0 and 24 points: Zero point corresponds to a person without complaints and the maximum value (24 points) to a patient with very severe limitations.
Quality of life (SF-36) | Baseline, endpoint (after 2 weeks) and the follow-up (after 1 month)
  The Medical Outcomes Short-Form Health Survey (SF-36) - a general health assessment instrument, originally created in English, which is easy to administer and understand. It consists of 36 questions, covering eight components, functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health assessed by 35 questions and one more comparative question between current and health one year ago.
Electrical activity of lumbar/multifidus (ML) and transverse abdominal (TrA) | Baseline, endpoint (after 2 weeks) and the follow-up (after 1 month)
  Surface Electromyography (EMGs) of the lumbar/multifidus (ML) and transverse abdominal (TrA) will be recorded using an 8-channel data acquisition system (model W4X8, Biometrics Ltd. , UK), bluetooth, with the following technical characteristics: hardware with 12-bit analog-to-digital (A/D) conversion board, 1000-fold gain amplifier, 20 to 500 Hz bandpass filter (2nd order Butterworth), common mode rejection ratio (RRMC) >100 dB, signal noise rate <3 mV RMS, 109 Ohms impedance, surface, bipolar, active, simple differential electrodes, 20-fold pre-amplification, reference electrode and DataLOG software for signal collection and analysis with 1000 Hz sampling frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraiba

IPD SHARING:
Plan to Share IPD: No